CLINICAL TRIAL: NCT02440243
Title: Grass Pollen Subcutaneous Immunotherapy: a Double-blind, Placebo-controlled Study in Elderly Patients With an Allergy to Grass Pollen
Brief Title: Grass Pollen Subcutaneous Immunotherapy in Elderly Patients
Acronym: SCITelderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Andrzej Bozek, Andrzej Bozek Assistant Professor, Director of Research, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC56871/12
Record Dates: First submitted 2015-04-22; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients active (Active Comparator): Purethal Grass
  Interventions: Drug: Purethal
- Patients placebo (Placebo Comparator): Placebo
  Interventions: Drug: Purethal -placebo

INTERVENTIONS:
Drug: Purethal — prerseasonal course of SCIT - three years
  Other Names: Vaccine
  Arms: Patients active
Drug: Purethal -placebo — preseasonal course of SCIT - three years
  Arms: Patients placebo

SUMMARY:
Background There is limited evidence indicating that specific immunotherapy in elderly patients is safe and effective. This study was performed to evaluate the safety and efficacy of specific subcutaneous immunotherapy (SCIT) against grass pollen allergens in patients over 60 years of age with seasonal allergic rhinitis (SAR) and a confirmed allergy to grass pollen.

Objective This study assessed the safety and efficacy of SCIT for grass pollen allergens in elderly patients with SAR.

Methods This study included 62 60- to 75-year-old patients with SAR and grass pollen allergy confirmed using a skin prick test, nasal provocation, and serum IgE measurement. The patients were individually randomized to the active or placebo groups using a double-blinded method. There were 33 subjects in the SCIT group (Purethal, Grass pollen, HAL Allergy B.V, Leiden, Netherlands) and 29 subjects in the placebo group monitored for three years. The patients were required to record each use of anti-allergy medication in a diary and use a visual graphic scale. The main outcome measure was the area under the curve (AUC) for the combined symptom and medication score (SMS).

DETAILED DESCRIPTION:
Methods Patients A total of 109 patients ranging from 60 to 70 years of age were recruited from the outpatient allergy clinic to assess their eligibility for inclusion in the study. The subjects had moderate or severe intermittent allergic rhinitis and fulfilled the ARIA criterion. Additionally, the patients included in the study all had a positive skin prick test (SPT), were positive for specific immunoglobulin E (sIgE), and had positive nasal provocation tests (NPTs) with grass pollen mixture allergens. Patients with any of the following characteristics were excluded from the study: hypersensitivity to other allergens, bronchial asthma, non-allergic rhinitis (especially senile or vasomotor rhinitis) and severe non-stable diseases. However, patients with stable coronary disease, diabetes, and arterial hypertension were permitted in the study. All subjects were required to abstain from anti-allergy drugs and glucocorticoid nasal drops for at least 6 weeks prior to the start of the study.

There were 62 patients individually randomized in comparable numbers to one of two "parallel" groups using a double-blind method. The groups were the active (n=33) treatment group and the placebo (n=29) group. There were 31 subjects in the SCIT group and 25 subjects in the placebo group that completed the three-year observation period. The groups were comparable at baseline.

Diagnostic procedures A careful examination of the eyes, ears, nose, and throat was performed on all patients. The severity of seasonal allergic rhinitis (SAR) was assessed using the Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines. The patients with other nasal problems such as chronic nasal obstruction, reduced olfaction, bacterial colonization, and chronic sinusitis were diagnosed based on a CT scan and nasal endoscopy. Several patients were excluded from further observation as a result of these problems. The subjects with other chronic or acute clinical disorders or with a history of respiratory tract infections within four weeks of the study initiation were also excluded. The SPT was performed using inhalant allergens (HAL Allergy B.V, Leiden, Netherlands) from the following panel: D. pteronyssinus, D. farinae, mixed 5 grasses (Phleum pratense, Dactylis glomerata, Anthoxanthum odoratum, Lolium perenne, and Poa pratensis), mixed tree, mugwort, Alternaria, Cladosporium, dog and cat allergens. There were also positive (10 mg/ml of histamine) and negative (saline) controls included. A grass pollen allergy was defined as having positive skin tests for 5 grass pollen allergens with a minimum wheal diameter of at least 3 mm greater than the negative control. The patients with negative tests for histamine sensitivity were excluded from further analyses. The sIgE reactivity to the single grass pollen allergen components (Phl p1, Phl p2, Phl p5, Phl p6, Phl p7 and Phl p12) was determined using ImmunoCAP (Phadia AB, Uppsala, Sweden) tests. The results were considered positive when the sIgE concentration was greater than 0.35 IU/ml (according to the manufacturer's instructions). NPTs were conducted using active anterior rhinomanometry with commercial grass pollen mixture allergens. The concentration was 10,000 AU/ml and the mixture was delivered as 1 puff per nostril (HAL Allergy B.V, Leiden, Netherlands) using the methods described by Bachert et al. and Dordal et al. A reduction in the peak nasal inspiratory flow greater than or equal to 40% and an increase in symptoms greater than or equal to 5 points were considered to be positive NPT criteria by Bachert et al. and Dordal et al. The NPTs were also repeated after three years of treatment. The patients monosensitized to grass pollen were included in this study.

Treatments The patients were randomly selected to receive Purethal Grasses 20,000 AUM/ml (pollen mixture extract solution of Agrostis stolonifera, Anthoxanthum odoratum, Arrhenatherum elatius, Dactylis glomerata, Festuca rubra, Holcus lanatus, Lolium perenne, Phleum pratense, Poa pratensis, Secale cereal, Loe edasi HAL Allergy B.V, Leiden, Netherlands) or placebo. The recruitment period was limited to three months (October-December). Purethal grasses (January-April) were administered as pre-seasonal therapy using the following regimen: 1 dose- 0.1 ml, 2 dose - 0.2 ml, 3 dose - 0.4 ml every week, and doses 4- 7 consisted of 0.5 ml every two weeks.

Using this schedule the average cumulative dose was 460,500 BAU (Bioequivalent Allergy Unit), which contains approximately 690 μg of Phl p5 administered to each patient undergoing active treatment for all three years of the study. The study consisted of two phases. The first phase was the baseline one season of follow-up visits without treatment and the second phase was three years of SCIT or placebo.

Assessment of efficacy The prime outcome measure was the area under the curve (AUC) for combined symptom and medication score (SMS) over the grass pollen season for baseline 2010 (before treatment) and in 2011, 2012 and finally in 2013 after three years of SCIT. The patients recorded symptom severity in a daily diary during the pollen season (May-August) by scoring the following areas: nasal itching, sneezing, running, blockage, and ocular itch on a separate Visual Analog Scale (VAS) with a continuous scale from 0 cm (no symptoms) to 10 cm (very severe symptoms). The rescue medication provided and scoring was a one point per spray for Azelastine nasal spray or eye drops (Levocabastine), or per 5 mg levocetirizine tablet. The score was two points per puff for mometasone fuorate nasal spray and three points per prednisolone 10 mg tablet. This combined symptom-medication score was calculated as a sum of the symptom score and medication score monitored daily with the use a diary as described. The SMS was derived by adding the VAS for each of these five symptoms.

The secondary outcome measures included quality of life, reduction of symptoms score, safety assessment and monitoring of IgG4. The local reactions were assessed at 30 min after injection and measured in cm. The systemic reactions were graded according to EAACI criteria.

Serum IgG4 measurements The serum concentration of IgG4 against birch alder and hazel pollens were determined in blood serum by ELISA tests according Lai et al. before and after the three-year SIT.

Quality of life Patient quality of life was evaluated with the RQLQ score for adults using questionnaires every grass pollen season during the study.

Pollen counts The local grass pollen counts were determined by volumetric pollen trap (Burkard, Scientific Ltd, Uxbridge, UK). The peak pollen count was defined as the day with highest grass pollen count for each season 3 weeks before and 3 weeks after the peak grass pollen count.

ELIGIBILITY:
Inclusion Criteria:

* a positive skin prick test (SPT), were positive for specific immunoglobulin E (sIgE), and had positive nasal provocation tests (NPTs) with grass pollen mixture allergens

Exclusion Criteria:

* hypersensitivity to other allergens, bronchial asthma, non-allergic rhinitis (especially senile or vasomotor rhinitis) and severe non-stable diseases.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The symptoms reduction as a compsite measure | three years
  The prime outcome measure was the area under the curve (AUC) for combined symptom and medication score (SMS)
Evaluation of symptomatic medication use reduction | three years
  Evaluation quantities of drugs based on patient diary.

SECONDARY OUTCOMES:
Number of patients with a local allergic reaction after injections | three years
  The local reactions were assessed at 30 min after injection and measured in cm.
Number of patients with a systemic allergic reaction after injections | three years
  The systemic reaction were assesed after injection according EAACI criteria.

REFERENCES:
- [Derived] Bozek A, Kolodziejczyk K, Krajewska-Wojtys A, Jarzab J. Pre-seasonal, subcutaneous immunotherapy: a double-blinded, placebo-controlled study in elderly patients with an allergy to grass. Ann Allergy Asthma Immunol. 2016 Feb;116(2):156-61. doi: 10.1016/j.anai.2015.12.013. PMID 26815709